CLINICAL TRIAL: NCT02114346
Title: Evaluating the Effect of High Dose Atorvastatin (80 mg/d) Comparing With Placebo in Preventing Contrast-induced Nephropathy in Patients Undergoing Computed Tomography Coronary Angiography
Brief Title: High Dose Atorvastatin for Preventing Contrast-induced Nephropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Hajian Nejad, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 392353
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Contrast-Induced Nephropathy
Keywords: Computed Tomography Angiogram; Side Effects; Contrast-Induced Nephropathy; Prevention
MeSH Terms: interventions — Atorvastatin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental): Patients in the atorvastatin group receive 80 mg atorvastatin (2 x atorvastatin 40 mg tablets) once daily from 24 hours before to 48 hours after administration of contrast material.
  Interventions: Drug: Atorvastatin; Drug: 0.9% sodium chloride
- Placebo (Placebo Comparator): Patients in the placebo group receive 2 placebo tablets once daily from 24 hours before to 48 hours after administration of contrast material.
  Interventions: Drug: Placebo; Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: Atorvastatin
  Arms: Atorvastatin
Drug: Placebo
  Arms: Placebo
Drug: 0.9% sodium chloride — Patients with estimated glomerular filtration rate of less than 60 mL/min/1.73 m2 are hydrated with 0.9% sodium chloride for 2 hours, from 1 hour before (3 mL/kg/hour) to 1 hour after (1 mL/kg/hour) operation. Patients with left ventricular ejection fraction less than 40% or New York Heart Association functional class III-IV, are hydrated with 0.5 mL/kg/hour.

SUMMARY:
The aim of this study is to determine the efficacy of atorvastatin in the prevention of contrast-induced nephropathy in patients undergoing computed tomography coronary angiography. Investigators assume that atorvastatin is effective in this regard. Investigators include patients referring for elective computed tomography coronary angiography and allocate them to atorvastatin or placebo from 24 hours before to 48 hours after administration of contrast material. Investigators then measure serum creatinine and see if it is raised by ≥ 0.5 mg/dL or ≥ 25% of the baseline value.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* candidate of elective computed tomography angiogram
* willingness to participate

Exclusion Criteria:

* unstable angina or myocardial infarction, cardiac arrhythmia, seizures, acute renal failure, end-stage renal disease
* unstable serum creatinine
* unstable hemodynamic
* intravascular administration of contrast material in the past month
* using high dose atorvastatin in the past month,
* known hypersensitivity to atorvastatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Plasma creatinine level | up to 48h after contrast injection
  Plasma creatinine level is measured at baseline and after 48 hours of contrast injection. Increase in plasma creatinine level ≥ 0.5 mg/dL or ≥ 25% of the baseline creatinine after 48 hours of contrast injection will be considered contrast induced nephropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Hajian, M.D., Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Alzahra Hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Li Y, Liu Y, Fu L, Mei C, Dai B. Efficacy of short-term high-dose statin in preventing contrast-induced nephropathy: a meta-analysis of seven randomized controlled trials. PLoS One. 2012;7(4):e34450. doi: 10.1371/journal.pone.0034450. Epub 2012 Apr 12. PMID 22511942